CLINICAL TRIAL: NCT03173729
Title: Point of Care, Real-time Urine Metabolomics Test to Diagnose Colorectal Cancers and Polyps in Low and Middle Income Countries
Brief Title: Point of Care Test to Diagnosed Colorectal Cancer and Polyps in Low Middle Income Countries
Status: Completed | Type: Observational
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, Olusegun Alatise, Dr, Obafemi Awolowo University Teaching Hospital
Other Study IDs: ERC/2017/02/11
Record Dates: First submitted 2017-05-23; First posted 2017-06-02 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A urine sample is collected with 3 weeks of their surgery or colonoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Phase 1 Cohort 1: CRC (n = 150)
- Phase 1 Cohort 2: Precancerous polyps (n = 150)
- Phase 1 Cohort 3: Normal controls (n = 150)
- Phase 2 Field Test: 75 patients who are high risk for CRC as described in the eligibility
  Interventions: Diagnostic Test: Biosensor Point of Care Device
- Phase 2 Validation Study Cohort 1: Family history of CRC (n = 330)
  Interventions: Diagnostic Test: Biosensor Point of Care Device
- Phase 2 Validation Study Cohort 2: LGI bleeding (n = 240)
  Interventions: Diagnostic Test: Biosensor Point of Care Device
- Phase 2 Validation Study Cohort 3: Patients with history of CRC (n = 75)
  Interventions: Diagnostic Test: Biosensor Point of Care Device

INTERVENTIONS:
Diagnostic Test: Biosensor Point of Care Device — This device is a point of care urine-based metabolomic diagnostic test that detects metabolite biomarkers for CRC and polyps.
  Groups: Phase 2 Field Test; Phase 2 Validation Study Cohort 1; Phase 2 Validation Study Cohort 2; Phase 2 Validation Study Cohort 3

SUMMARY:
This is a-two phase study. Phase 1 will adapt a 3-metabolite biosensor that identifies patients with colorectal cancer (CRC) and precancerous polyps to Nigerian patients. Phase 2 will pilot test and evaluate the point-of-care (POC) biosensor device in Nigeria.

DETAILED DESCRIPTION:
In Phase 1, urine will be collected from 450 Nigerian patients (150 with CRC, 150 with polyps, and 150 patients with no colon premalignant or malignant pathology. These samples will be used to refine a handheld biosensor. This handheld biosensor is intended to be a cost-effective POC diagnostic test highly sensitive for CRC in Nigerian patients.

In Phase 2, the biosensor device will be piloted in Nigeria with 75 patients that are high-risk for CRC.. After the pilot, POC test in real-time analysis on urine from 645 patients who are in one of three groups: 1.> 40 years of age with rectal bleeding; 2.a family history of CRC; 3. have a diagnosis of CRC. All patients will receive a colonoscopy. Beliefs and barriers related to urine testing for CRC will be investigated. Study will be completed within 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 40 years of age with LGI bleeding OR
* Patients who are high risk due to family history of CRC

  o Must be at most 10 years younger than when relative presented with CRC (for example, a patient with a relative diagnosed at age 40 with CRC will be eligible after age 30) OR
* Patients with a diagnosis of stage I-III CRC who have no evidence of disease

Exclusion Criteria:

* Patients who are unable to provide written informed consent;
* Previous diagnosis, treatment, or surgery for any cancer other than CRC
* Age younger than 40 years with no family history of CRC
* Any significant medical comorbidities
* Inability to provide a urine sample no fewer than 3 days before colonoscopy
* Inability to fully complete the patient satisfaction survey tool
* Diagnosis of or suspected inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in Phase 1 has a pathologic diagnosis of colon cancer (either by colonoscopy or resection specimens), or colonoscopy demonstrating adenomatous polyps or no colon premalignant or malignant pathology.
  Patients in Phase 2 are > 40 years of age with LGI bleeding, or at high-risk due to family history, or with a history of CRC
Sampling Method: Non-Probability Sample
Enrollment: 926 (Actual)
Dates: Start 2017-02-11 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of a point of care device to diagnose colorectal cancer and polyps | 5 years
  We have designed a urine-based point of care diagnostic test to risk-stratify patients at high-risk for colorectal cancer. that will have 50% specificity and 80% sensitivity among Nigerian targeted population.

SECONDARY OUTCOMES:
Number of patients that are willing to consider continued colorectal cancer surveillance with a urine point of care test. | 3 years
  The barriers and attitudes of patients towards a point of care urine test will be used to predict how many patients are willing to use this methodology.
Cost per patient of point of care urine test for diagnosing patients with colorectal cancer and polyps. | 3 years
  The cost per patient will be determined using a cost effectiveness model already developed for the urine screening test in high-income countries.

CONTACTS AND LOCATIONS:
Locations (5):
- Nigeria (5):
  - Endoscopy Unit, University of Ilorin Teaching Hospital, Ilorin, Kwara State
  - Federal Medical Center, Owo, Ondo State
  - Endoscopy Unit, University College Hospital, Ibadan, Osun State
  - Endoscopy Unit, Obafemi Awolowo University Teaching Hospitals, Ile-Ife, Osun State
  - Ladoke Akintola University Teaching Hospital, Osogbo, Osun State

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH/NCI approved guidelines